CLINICAL TRIAL: NCT00272168
Title: The Use of Skills Training to Augment CWT/VI for Veterans With SMI
Brief Title: The Use of Skills Training to Augment Compensated Work Therapy (CWT)/VI for Veterans With SMI
Acronym: MPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3437-R; H-26250 (Other: University of Maryland, Baltimore IRB number)
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Mental Illness; Schizophrenia
Keywords: Cognitive behavioral therapy; Social Skills training; Vocational Rehabilitation
MeSH Terms: conditions — Mental Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: MPROVE (Experimental): The Maryland Program for Vocational Effectiveness (MPROVE)
  Interventions: Behavioral: Maryland Program for Vocational Effectiveness
- Arm 2: Control (Active Comparator): Supportive Treatment for SMI (control)
  Interventions: Other: Supportive Treatment for SMI

INTERVENTIONS:
Behavioral: Maryland Program for Vocational Effectiveness — psychosocial intervention that combines elements of cognitive-behavioral therapy (CBT) with work-related social skills training and basic problem solving training (SST)
  Other Names: M-PROVE
  Arms: Arm 1: MPROVE
Other: Supportive Treatment for SMI — Sessions are interactive, supportive, flexible, and unstructured, and are intended to help patients adjust to their new jobs and understand how working affects their lives. The therapist stance is non-directive, and there is an emphasis on having patients share with one another, rather than having the therapists dictate the content of group sessions. The primary goals of the therapists are to engage patients in treatment and to generate discussion among members.
  Other Names: STS
  Arms: Arm 2: Control

SUMMARY:
The goal of this study is to evaluate the efficacy of a combined social skills training and cognitive-behavioral therapy intervention for seriously mentally ill Veterans as they begin employment.

DETAILED DESCRIPTION:
In spite of the fact that most individuals with serious mental illness (SMI) express a desire to work, some 80% of these individuals in the United States are chronically unemployed or under-employed. The VA has long recognized the need for vocational rehabilitation programs to facilitate meaningful work for patents with SMI. VA vocational rehabilitation programs (Compensated Work Therapy / Veterans Industries; CWT/VI) generally follow a supported employment model which has been the most extensively studied type of program and has garnered the most empirical support for helping individuals with SMI obtain employment. Nevertheless, studies of supported employment programs find that approximately 50% of participants remain unemployed and that job retention rates among those patients who do get jobs are quite low. In fact, more than half of all clients leave their supported employment positions within 6 months. The most frequently cited reasons for job terminations among patients with SMI include interpersonal problems in the work place and difficulty coping with symptom exacerbations.

The investigators have developed a psychosocial intervention (CBT-SST) that is designed to augment CWT/VI by targeting the skills needed for reintegration into community work settings and to facilitate job retention among persons with SMI. It is a manualized intervention that combines elements of cognitive-behavioral therapy (CBT) with work-related social skills training and basic problem solving training (SST). The CBT module of the treatment is designed to help reduce residual symptoms of mental illness and help patients develop strategies to cope with symptom exacerbations when they occur. The SST social skills and problem solving modules are designed to help patients improve their interpersonal functioning at work.

The purpose of this study is to conduct a randomized clinical trial comparing CWT/VI augmented with CBT-SST to CWT/VI without augmentation (control condition). The investigators will recruit patients for the study as they are beginning jobs through enrollment in the CWT/VI program at the VA, as this is the critical time period for them to develop the skills needed to perform well and retain employment. Expected outcomes for CBT-SST participants relative to controls include improved job retention and earnings, improved social skills (as assessed both in the clinic and in the actual work place), better everyday problem solving skills / social function, and improvements in quality of life.

The long term objective of this research is to develop and disseminate an effective skills training program that can improve work function and job retention among persons with SMI, and thereby enhance: a) their social role functioning; and b) their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder, or other severe mental disorder including bipolar disorder, major depression, or severe anxiety disorder
* Enrolled in vocational rehabilitation program or working
* Age between 18 and 65 years
* Ability and willingness to attend treatment sessions for 3 months
* Judged by their treating clinician to be able to participate and provide informed consent
* Ability and willingness to provide informed consent to participate

Exclusion Criteria:

* Documented history of severe neurological disorder or head trauma with ongoing cognitive sequelae
* Inability to effectively participate in the baseline assessments due to intoxication or psychiatric symptoms on two successive appointments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Tenhula, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2: Control: Supportive Treatment for Serious Mental Illness (control)
  Supportive Treatment for Serious Mental Illness (SMI): Sessions are interactive, supportive, flexible, and unstructured, and are intended to help patients adjust to their new jobs and understand how working affects their lives. The therapist stance is non-directive, and there is an emphasis on having patients share with one another, rather than having the therapists dictate the content of group sessions. The primary goals of the therapists are to engage patients in treatment and to generate discussion among members.
Period: Overall Study
Arm/Group | Arm 1: MPROVE | Arm 2: Control
Started | 47 | 41
Completed | 37 | 31
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: MPROVE | Arm 2: Control | Total
Number analyzed (Participants) | 47 | 41 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.47 (6.29) | 51.51 (6.07) | 51.49 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 34 | 73
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 47 | 41 | 88

OUTCOME MEASURES:

1. Primary Outcome: Employment Status
Description: Data collected included from participants: 1) hours scheduled to work per week and 2) weekly wages earned.
Time Frame: Post Treatment (approximately 3 months after completion of the baseline assessment)
Measure: Mean (Standard Deviation); unit: Hours worked per week
Arm/Group | Arm 1: MPROVE | Arm 2: Control
Number analyzed (Participants) | 37 | 31
Hours worked per week | 26.2 (12.39) | 24.83 (9.43)

2. Secondary Outcome: Cognitive Insight
Description: Cognitive insight was assessed using the Beck Cognitive Insight Scale, a 15-item questionnaire developed to evaluate patients' self-reflectiveness and their overconfidence in their interpretations of their experiences. Participant responses to each of these items were as follows:
  1. Do not agree at all
  2. Agree slightly
  3. Agree a lot
  4. Agree completely
  Total score for the self-certainty scale could range from 6 to 24. Total score for the self-reflectiveness scale could range from 9 to 36. Total score for the composite score was calculated by subtracting the summed score for the self-certainty scale from the summed score of the self-reflectiveness scale and could range from 3 to 12, lower composite scores are an indicator of lower psychiatric functioning.
Time Frame: Post Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: MPROVE | Arm 2: Control
Number analyzed (Participants) | 37 | 31
units on a scale | 9.56 (5.32) | 7.29 (5.79)

3. Secondary Outcome: Psychiatric Symptoms
Description: Psychiatric Symptoms were assessed using the Brief Psychiatric Rating Scale (BPRS), a widely used instrument for assessing the positive, negative, and affective symptoms of individuals who have mental illnesses. The BPRS consists of 20 symptom constructs scored from 1 (not present) to 7 (extremely severe). BPRS total score could range from 0 (not present) to 140 (extremely severe).
Time Frame: Post-Treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: MPROVE | Arm 2: Control
Number analyzed (Participants) | 47 | 41
scores on a scale | 36.25 (8.69) | 38.71 (10.63)

4. Primary Outcome: Work Performance (Work Behavior Inventory)
Description: This measure is completed with participants' supervisors and assesses current work behavior and vocational function. The WBI yields six scores related to fundamental work requirements: social skills, cooperativeness, work habits, work quality personal presentation, and a general score of overall work performance. Each of these is rated between 1-5:
  1. Consistently an area Needing Improvement
  2. Occasionally an area Needing Improvement
  3. Performance Adequate in this area
  4. Occasionally an area of Superior Performance
  5. Consistently an area of Superior Performance.
  The global impression of work behavior (overall rating of work functioning using the same 1-5 scale) was used for the purpose of reporting results for this study.
Time Frame: Post Treatment
Measure: Mean (Standard Deviation); unit: rating on a scale
Arm/Group | Arm 1: MPROVE | Arm 2: Control
Number analyzed (Participants) | 37 | 31
rating on a scale | 2.37 (0.76) | 2.37 (0.74)

5. Primary Outcome: Social Functioning
Description: This was assessed using the Maryland Assessment of Social Competence (MASC), which assesses participants social problem solving skill abilities in both work-related and non-work related situations. Using three scenes, the participant is rated on the following scale for each scene. Overall score is then averaged to arrive at a final score.
  1. Very Poor
  2. Poor
  3. Neither good nor poor
  4. Somewhat good
  5. Very good
Time Frame: Post Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: MPROVE | Arm 2: Control
Number analyzed (Participants) | 37 | 31
units on a scale | 3.69 (1.2) | 3.56 (1.31)

6. Primary Outcome: Employment Status
Description: Data collected included from participants: weekly wages earned
Time Frame: Post Treatment (approximately 3 months after completion of the baseline assessment)
Measure: Mean (Standard Deviation); unit: dollars/week
Arm/Group | Arm 1: MPROVE | Arm 2: Control
Number analyzed (Participants) | 37 | 31
dollars/week | 143.08 (186.76) | 72.07 (79.81)

ADVERSE EVENTS:
Time Frame: Duration of participants involvement in the study, which was approximately 12 months.
Arm/Group | Arm 1: MPROVE | Arm 2: Control
Serious Adverse Events (participants affected / at risk) | 13/47 | 9/41
Other Adverse Events (participants affected / at risk) | 0/47 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: MPROVE (N=47) | Arm 2: Control (N=41)
Medical Hospitalization (General disorders) | 7 | 2
Psychiatric Hospitalization (Psychiatric disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No